CLINICAL TRIAL: NCT05677672
Title: Phase I/Ⅱ Study to Evaluate the Safety and Efficacy of Human TH-SC01 Cell Injection in the Treatment of Complex Perianal Fistula
Brief Title: The Purpose of This Study is to Evaluate the Safety and Efficacy of Human TH-SC01 Cell Injection in the Treatment of Complex Perianal Fistula
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Topcel-KH Pharmaceutical Co., Ltd. (Industry)
Collaborators: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TH-SC01-CAF-Ⅰ/Ⅱ 1.0
Record Dates: First submitted 2022-12-14; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Complex Perianal Fistulas
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Phase 1 was a non-randomized, single-arm, multicenter, dose-escalation clinical trial design.
  Phase 2 was a randomized, double-masking , multicenter, blank control, dose-extended clinical trial design.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human TH-SC01 cell injection (Experimental): Human TH-SC01 Cell Injection is a human expanded umbilical cord mesenchymal stem cells suspension
  Interventions: Biological: Human TH-SC01 Cell Injection
- Placebo-control group (Placebo Comparator): Saline solution
  Interventions: Other: Saline solution

INTERVENTIONS:
Biological: Human TH-SC01 Cell Injection — Single injection of 0.6×10^7,1.2×10^8, 1.8×10^8 cells/kg
  Arms: Human TH-SC01 cell injection
Other: Saline solution — saline solution will be given at the same quantity and following the same schedule
  Arms: Placebo-control group

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of human TH-SC01 cell injection for the treatment of complex perianal fistulas

DETAILED DESCRIPTION:
This study is a phase Ⅰ/Ⅱ study, Phase 1 was the dose increment phase, and phase 2 was the expansion phase

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Subjects aged between 18 and 70, both male and female.
3. The subject was clinically diagnosed as complex anal fistula. The diagnostic criteria for complex anal fistula were adopted by the 2016 American Association of Colorectal Surgeons Guidelines for the Treatment of Perianal Abscess, Anal Fistula and Rectovaginal Fistula.
4. The subjects had received conventional treatment for anal fistulas
5. All subjects and their partners were not planning to have a child from screening to the end of the trial and agreed to use effective non-drug contraception during the trial.

Exclusion Criteria:

1. Subjects with anal fistula in the acute infection period.
2. Subjects with abscess or collections >2 cm.
3. Subjects with abnormal laboratory results: liver function: total bilirubin >=1.5 × ULN, and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >=2 × ULN; renal function: creatinine clearance below 60 mL/minute calculated using Cockcroft-Gault formula or by serum creatinine >=1.5 × upper limit of normal (ULN).
4. Subjects with malignant tumors or a history of malignant tumors.
5. Subjects with severe, progressive, uncontrolled hepatic, hematological, gastrointestinal (except Crohn's disease), endocrine, pulmonary, cardiac, neurological, psychiatric, or cerebral diseases.
6. Serum virology test (HBeAg, HCV antibody, HIV antibody, Treponema pallidum antibody) positive.
7. Subjects allergic to gentamicin sulfate, anesthetics or contrast media.
8. Subjects allergic to MRI contrast.
9. Subjects who has major surgery or severe trauma within 6 months prior to the screening period.
10. Subjects who has received any investigational drug within 3 months prior to the screening.
11. Subjects deemed inappropriate by the investigator to participate in this clinical trial.
12. The female participant who is pregnant, or is lactating.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-12-30 (Estimated); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Severity and incidence of study drug-related adverse-events | Day 28 (Week 4)
  Severity and incidence of study drug-related adverse-events within D28(W4) after administration.
Dose-limiting toxicity (DLT) | Day 28
  Exploration of dose-limiting toxicity (DLT)
maximum tolerated dose (MTD) | Day 28
  Exploration of maximum tolerated dose(MTD)
Percentage of effectiveness | Day 84
  Percentage of effectiveness at 84 days of administration by MRI imaging evaluated fistula healing with no or minimal effusion

SECONDARY OUTCOMES:
Severity and incidence of study drug-related adverse-events | Day 28
  Severity and incidence of study drug-related adverse-events after D28(W4) after administration.

OTHER OUTCOMES:
Patient quality of life score | Week 1-Week 52
  Change from baseline in Patient quality of life score from W1-W52
Rate of recurrence | Week 24-Week 104
  The recurrence rate after administration
Closure time of fistulas | Day 1
  Closure time of wound and fistula at the anal fistula surgical site after drug administration: Starting from the next day after administration (D1).
SF-36 score | Week 1-Week 52
  Change From Baseline in SF-36 score after administration，
Van Assche Score | Day 0-Week 52
  Change From Baseline in Van Assche Score.Total score ranges from 0 to 10. Higher score means more pain.
Wexner incontinence Score | Week 4-Week 52
  Change From Baseline in Wexner incontinence Score .Total score ranges from 0 to 20. Higher score means more severe disease.
Anal sphincter function： rectal pressure | Week 4-Week 52
  Change from baseline in rectal pressure，In healthy people, the pressure ranges from 60 to 150mmHg, with the internal sphincter pressure accounts for about 80% and external sphincter pressure accounts for 20%.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital Central University, Changsha, Hunan, China